CLINICAL TRIAL: NCT01567280
Title: International Cross-sectional and Longitudinal Assessment on Asthma Control (Liaison)
Acronym: LIAISON
Status: Completed | Type: Observational
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: DFIDM-1101
Record Dates: First submitted 2012-03-29; First posted 2012-03-30 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Controlled patients: Asthmatic patients with controlled asthma (according to ACQ score)
- Partly controlled/Uncontrolled patients: Patients with partly controlled or uncontrolled asthma (according to ACQ score)

SUMMARY:
The study design consists of a cross-sectional survey on the clinical characteristics of patients with asthma and their level of asthma control and current quality of life, and on a prospective evaluation of the rate of switch from the uncontrolled/poorly controlled condition to the status of controlled asthma. Asthma control will be based on the Asthma Control Questionnaire scoring system, that has been fully validated for use in both clinical practice and clinical trials and has strong discriminative properties which means that it can detect small differences between patients with different levels of asthma control and it is very sensitive to within-patient change in asthma control over time.

Quality of life as a reflection of the control of the disease, will also be evaluated by means of the Mini Asthma Quality of Life Questionnaire scoring system.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. Written informed consent obtained.
  2. Male or female adult (at least 18 years of age) patients with asthma diagnosed (according to GINA guidelines and confirmed by a chest physician) for at least 6 months.
  3. Patients in treatment with the same antiasthmatic drugs in the last 4 weeks before enrolment.
* Exclusion criteria:

  1. Patients enrolled in clinical trial in the previous 4 weeks or subjects already admitted in this study.
  2. Patients suffering from conditions and illnesses that might interfere with the study purpose, according to the investigator's evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthmatic patients (in treatment with the same antiasthmatic therapy for at least 4 weeks) visiting the centre.
Sampling Method: Probability Sample
Enrollment: 8111 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Asthma Control Questionnaire score | 3 months
Mini Asthma Quality of Life Questionnaire score | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Sanitaria Firenze Piero Palagi, Florence, Italy

REFERENCES:
- [Background] Braido F, Brusselle G, Ingrassia E, Nicolini G, Price D, Roche N, Soriano JB, Worth H; LIAISON study group. InternationaL cross-sectIonAl and longItudinal assessment on aSthma cONtrol in European adult patients--the LIAISON study protocol. BMC Pulm Med. 2013 Mar 25;13:18. doi: 10.1186/1471-2466-13-18. PMID 23530817
- [Result] Braido F, Brusselle G, Guastalla D, Ingrassia E, Nicolini G, Price D, Roche N, Soriano JB, Worth H; LIAISON Study Group. Determinants and impact of suboptimal asthma control in Europe: The INTERNATIONAL CROSS-SECTIONAL AND LONGITUDINAL ASSESSMENT ON ASTHMA CONTROL (LIAISON) study. Respir Res. 2016 May 14;17(1):51. doi: 10.1186/s12931-016-0374-z. PMID 27179604